CLINICAL TRIAL: NCT04224311
Title: Immunogenicity of Quadrivalent Meningococcal Conjugate Vaccine in Frequent Platelets Donors
Acronym: PLAT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lindsey R. Baden, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019P003638
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Preventive Immunization; Meningitis
MeSH Terms: conditions — Meningitis | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low number plateletpheresis donations (Active Comparator): Participants that have had 1-2 plateletpheresis donations in the last 365 days. Menactra will be administered as a 0.5 mL dose.
  Interventions: Biological: Menactra
- Medium number plateletpheresis donations (Active Comparator): Participants that have had 3-19 plateletpheresis donations in the last 365 days. Menactra will be administered as a 0.5 mL dose.
  Interventions: Biological: Menactra
- High number plateletpheresis donations (Active Comparator): Participants that have had 20-24 plateletpheresis donations in the last 365 days. Menactra will be administered as a 0.5 mL dose.
  Interventions: Biological: Menactra

INTERVENTIONS:
Biological: Menactra — 0.5 mL dosage of Menactra will be administered by intramuscular injection in the deltoid muscle on day 0.

SUMMARY:
In this study, the investigators will evaluate the immunogenicity of a quadrivalent conjugate meningococcal vaccine in healthy, plateletpheresis donors.

DETAILED DESCRIPTION:
This will be an open-label prospective vaccine response study evaluating one dose of MenACWY-D in plateletpheresis donors at the Brigham and Women's Hospital (BWH). Potential participants will be divided into three groups according to the number of plateletpheresis within 365 days of enrollment (including the day of enrollment): 1-2 sessions group (considered as the control group), 3-19 sessions group, 20-24 sessions group and randomly sampled from in allocation proportions of 0.45, 0.10, and 0.45, respectively; justification for this approach is provided in the Statistical Analysis section. MenACWY-D vaccine will be administered to each patient. Pre- and post-vaccination blood will be collected to assess immunogenicity, likely using serum bactericidal antibody (SBA) against Neisseria meningitidis for each serogroup. Immunogenicity will be primarily evaluated by seroresponse such as a fourfold increase of SBA titers between pre- and post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years old or older
* Meet the standard requirements to donate platelets
* Have had at least one plateletpheresis in the prior 365 days (including the day of enrollment)

Exclusion Criteria:

* Participants who donated platelets in any other medical center in the previous 365 days
* Severe allergic reaction to a previous meningococcal vaccine or to any component of MenACYW-D
* History of Guillain-Barré syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Seroresponse of vaccine | Months 1 and 6.
  The primary outcome will be the seroresponse of MenACYW-D vaccination, such as a fourfold change of SBA titers between pre- and post-vaccination for each of the 4 antigens.

SECONDARY OUTCOMES:
Seroprotection | Months 1 and 6.
  The pre- and post-vaccination seroprotection, such as SBA titer greater than or equal to 1:8.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Baden, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available upon request to the principal investigator following the publication of the primary manuscript.

REFERENCES:
- [Derived] Desjardins M, Cunningham P, Mitre X, Pierre D, Montesano C, Woods T, Oganezova K, Krauss JH, Von SS, Kupelian JA, Li X, Gothing JA, Kleinjan JA, Zhou G, Piantadosi S, Sherman AC, Walsh SR, Issa NC, Kaufman RM, Baden LR. Immunogenicity of quadrivalent meningococcal conjugate vaccine in frequent platelet donors. Blood. 2023 Jul 13;142(2):202-209. doi: 10.1182/blood.2022019482. PMID 37172200